CLINICAL TRIAL: NCT03869450
Title: A Multi-center, Evaluator-blinded Study to Evaluate Effectiveness and Safety of HA Fillers for Lifting, Contouring and Correcting Volume Deficiency of the Midface Using an Individualized Treatment Algorithm
Brief Title: A Study to Evaluate Effectiveness and Safety of Hyaluronic Acid (HA) Fillers
Acronym: 05DF1707
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05DF1707
Record Dates: First submitted 2018-11-14; First posted 2019-03-11 (Actual); Results first posted 2020-04-02 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2020-04

CONDITIONS: Volume Deficiency of the Midface

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Restylane Volyme (Experimental): According to the treatment algorithm, treated with Restylane Volyme
  Interventions: Device: Restylane Volyme
- Restylane Defyne (Experimental): According to the treatment algorithm, treated with Restylane Defyne
  Interventions: Device: Restylane Defyne
- Restylane Lyft Lidocaine (Experimental): According to the treatment algorithm, treated with Restylane Lyft Lidocaine
  Interventions: Device: Restylane Lyft Lidocaine

INTERVENTIONS:
Device: Restylane Volyme — Hyaluronic based filler
  Arms: Restylane Volyme
Device: Restylane Defyne — Hyaluronic based filler
  Arms: Restylane Defyne
Device: Restylane Lyft Lidocaine — Hyaluronic based filler
  Arms: Restylane Lyft Lidocaine

SUMMARY:
The purpose of the study is to investigate the degree of improvement in appearance after treatment with different hyaluronic acid (HA) fillers. Product selection is based on Investigator assessment of participant tissue coverage and main treatment goal (volumizing, lifting or contouring).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female 25 to 55 years old that needs lifting, contouring or volumization of the midface
* Signed and dated informed consent

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel and lidocain
* Previous use of any permanent or semi-permanent facial tissue augmentation therapy or contouring with, lifting threads, permanent implants, or autologous fat in the treatment area
* Previous use of any HA or collagen based facial tissue augmentation therapy in the facial area, any previous use of neurotoxin or any previous facial surgery
* Any medical condition that in the opinion of the Investigator would make the participant unsuitable for inclusion

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (3):
- Galderma Research Site, Munich, Germany
- Galderma Research Site, Palermo, Italy
- Galderma Research Site, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Volyme | Restylane Defyne | Restylane Lyft Lidocaine
Started | 31 | 25 | 34
Completed | 30 | 23 | 34
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Restylane Volyme: According to the treatment algorithm, Restylane Volyme was chosen for participants whose primary need for treatment was volume deficiency.
  Restylane Volyme: Hyaluronic based filler
- Restylane Defyne: According to the treatment algorithm, Restylane Defyne was chosen for participants with thin tissue coverage and whose primary need for treatment was lifting or contouring.
  Restylane Defyne: Hyaluronic based filler
- Restylane Lyft Lidocaine: According to the treatment algorithm, Restylane Lyft Lidocaine was chosen for participants with thick tissue coverage and whose primary need for treatment was lifting or contouring.
  Restylane Lyft Lidocaine: Hyaluronic based filler
- Total: Total of all reporting groups
Arm/Group | Restylane Volyme | Restylane Defyne | Restylane Lyft Lidocaine | Total
Number analyzed (Participants) | 31 | 25 | 34 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 25 | 34 | 90
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 29 | 74
  Male | 5 | 6 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 31 | 24 | 34 | 89
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 10 | 7 | 13 | 30
  United Kingdom | 10 | 10 | 10 | 30
  Germany | 11 | 8 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Aesthetic Improvement of Midface
Description: A blinded evaluator assesses the improvement compared to baseline (pre-treatment) using a 5-graded scale; Worse, No change, Improved, Much improved or Very much improved. Aesthetic improvement of midface is defined as those participants assessed as Improved, Much improved or Very much improved.
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane Volyme | Restylane Defyne | Restylane Lyft Lidocaine
Number analyzed (Participants) | 31 | 24 | 34
percentage of participants | 96.8 [83.3 to 99.9] | 100 [85.8 to 100.0] | 97.1 [84.7 to 99.9]

2. Secondary Outcome: Percentage of Participants With Improved Midface Volume
Description: A blinded evaluator assessed the fullness of the midface by using a 4-graded scale where 1= fairly full and 4= substantial loss of fullness.
  Improved midface volume was defined as at least a 1-grade decrease from baseline.
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Restylane Volyme | Restylane Defyne | Restylane Lyft Lidocaine
Number analyzed (Participants) | 31 | 24 | 34
percentage of participants | 90.3 [74.2 to 98.0] | 87.5 [67.6 to 97.3] | 79.4 [62.1 to 91.3]

3. Secondary Outcome: Percentage of Participants Assessed as Having Natural Treatment Results
Description: Blinded evaluator assessed participants by answering Strongly agree/Agree/Neither agree nor disagree/Disagree/Strongly disagree to the question "Are the subject's treatment results natural looking?". Having natural treatment results is defined as being assessed with answers Strongly agree or Agree.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Volyme | Restylane Defyne | Restylane Lyft Lidocaine
Number analyzed (Participants) | 31 | 24 | 33
percentage of participants | 93.5 | 100 | 93.9

ADVERSE EVENTS:
Time Frame: 24-27 weeks (depending on how long screening period), from signature of informed consent to last study visit.
Arm/Group | Restylane Volyme | Restylane Defyne | Restylane Lyft Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/25 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/25 | 0/34
Other Adverse Events (participants affected / at risk) | 3/31 | 0/25 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Volyme (N=31) | Restylane Defyne (N=25) | Restylane Lyft Lidocaine (N=34)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) — Not related to study product or injection procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03869450/Prot_SAP_000.pdf